CLINICAL TRIAL: NCT05030194
Title: Comparing Nicotine Delivery, Subjective Effects, and Sensory Experiences of Tobacco Users Using Oral Nicotine Products and Electronic Cigarettes [ZYN Study]
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: I 1574221
Record Dates: First submitted 2021-08-30; First posted 2021-09-01 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Tobacco Use; Tobacco Smoking; Cigarette Smoking; Smokeless Tobacco Cessation
MeSH Terms: conditions — Tobacco Use; Tobacco Smoking; Cigarette Smoking; Tobacco Use Cessation | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Order 1 - Oral Nicotine product - ZYN and Electronic Cigarettes (Experimental): Participants will use each product for up to a 30 minute interval But will also be permitted to stop use before the end of the 30-minute ad lib use period
  Interventions: Other: Electronic Cigarette; Other: Oral Nicotine Pouch
- Order 2 - Electronic Cigarettes and Oral Nicotine product (Experimental): Participants will use each prodcut for up to 30 minutes but will also be permitted to stop use before the end of the 30-minute ad lib use period
  Interventions: Other: Electronic Cigarette; Other: Oral Nicotine Pouch

INTERVENTIONS:
Other: Electronic Cigarette — Participants engage in 30 minutes of an oral nicotine product. In those 30 minutes the product can be used as much or as little as preferred.
  Other Names: Vuse Alto
Other: Oral Nicotine Pouch — Participants will be instructed to place a 6mg nicotine pouch in their mouth between gum and lip for up to 30 minutes.
  Other Names: ZYN

SUMMARY:
To pilot test the appeal of non-tobacco oral nicotine products in cigarette smokers, smokeless tobacco users, and oral nicotine users.

DETAILED DESCRIPTION:
This study will assess the use, nicotine delivery, subjective response, and sensory appeal of an oral nicotine product (ZYN) compared to electronic nicotine delivery systems (ENDS, Vuse Alto) in cigarette smokers, smokeless tobacco users and oral nicotine users.

ELIGIBILITY:
Inclusion Criteria:

* Current daily cigarette smoker as determined by:

  1. Smokes >5 cigarettes/day for >1 year OR
  2. Current daily smokeless tobacco or oral nicotine user as determined by:

  a. Uses >=5 units/day for >=1 year
* b. Uses portioned moist snuff, loose moist snuff and/or nicotine patches
* Willingness to abstain from using cigarettes/ST (smokeless tobacco) for 8-10 hours (overnight abstinence) prior to study visits (verified by exhaled-air carbon monoxide < 10ppm).
* Self-report fair or better physical health.
* Self-report fair or better mental health.
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related products

Exclusion Criteria:

* Currently uses other tobacco or nicotine products (e.g., ENDS) > 2 days/week.
* Self-report having active, untreated medical/psychiatric conditions History of serious side effects from nicotine or from any nicotine replacement therapies.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Nursing female participants.
* Vulnerable populations, such as cognitively impaired adults, individuals who are not yet adults, pregnant women, and prisoners.
* Unwilling or unable to follow protocol requirements.
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive study drug.
* Previous use of the study products (ZYN or Vuse Alto; on! or General Slims).

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Change in nicotine boost | up to week 4
  will be measured as the post bout plasma nicotine concentration minus the pre-bout plasma nicotine concentration
Change in sensory response | up to 1 year
  will be measured by a Questionnaire scored on a 0-100 visual analog scale with 0 (Not at all) to 100 (Extremely).

SECONDARY OUTCOMES:
Change is stress markers | Up to 4 weeks
  Saliva will be collected before and after product use of each product to establish plasma nicotine concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Goniewicz, PhD, Principal Investigator — Roswell Park Comprehensive Cancer Center
Locations (1):
- Roswell Park Comprehensive Cancer Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No